CLINICAL TRIAL: NCT01073345
Title: Portal Venous Hemodynamic Changes After Hepatectomy and the Incidence of Postoperative Ascites
Brief Title: Portal Venous Hemodynamic Changes After Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. Jürgen Weitz, MSc, University of Heidelberg
Other Study IDs: NNR-4
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Ascites; Hepatectomy
Keywords: Patients undergoing elective hepatic resection
MeSH Terms: conditions — Ascites | interventions — Portal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for liver function tests and cytokine levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Major hepatic resection: Patients undergoing resection of > 2 liver segments
  Interventions: Procedure: Portal venous pressure; Procedure: Portal venous flow; Procedure: Hepatic artery flow
- Minor hepatic resection: Patients undergoing resection of </= 2 liver segments
  Interventions: Procedure: Portal venous pressure; Procedure: Portal venous flow; Procedure: Hepatic artery flow
- Control group: Patients undergoing exploratory laparotomy for hepatobiliary disease without resection (e.g. due to inoperable disease)
  Interventions: Procedure: Portal venous pressure; Procedure: Portal venous flow; Procedure: Hepatic artery flow

INTERVENTIONS:
Procedure: Portal venous pressure — Portal venous pressure is measured by invasive means using an arterial canula
Procedure: Portal venous flow — Portal venous flow is measures using a noninvasive method (Doppler flow meter)
Procedure: Hepatic artery flow — Hepatic artery flow will be measured using a noninvasive method (Doppler flow meter)

SUMMARY:
The aim of this study is to investigate the pathophysiological mechanisms underlying the formation of posthepatectomy ascites with a focus on the significance of changes in portal venous hemodynamics after hepatic resection. By evaluation of other factors that may be involved in the formation of ascites this study may help to show to what extent the increase of portal venous pressure contributes to ascites formation. Detailed knowledge about pathogenetic factors concerning the formation of postoperative ascites might help preventing protracted hospital stay and further inconveniences to the patient.

DETAILED DESCRIPTION:
The mechanisms underlying the development of large-volume ascites after hepatectomy remain poorly understood. While studies on animal models suggest an increase of portal venous pressure after hepatectomy that may in turn favor the transudation of fluid into the peritoneal cavity further factors may be critically involved in the postoperative formation of ascites. These factors may include a drop in serum protein levels (and colloid osmotic pressure), a transient impairment in renal function and a surgery-induced capillary leakage. However, a better knowledge of the pathophysiology represents the prerequisite for efficient treatment.

In the present study the impact of changes in hepatic hemodynamics after hepatectomy on development of ascites will be investigated. Enrolled patients will receive measurement of portal venous flow and pressure as well as hepatic artery flow before and after hepatic resection. Associations of changes in these parameters with development of postoperative ascites and further postoperative complications will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective hepatic resection
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Evidence of ascites or hypalbuminemia preoperatively
* Renal insufficiency
* Expected lack of compliance
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at a University Hospital
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative ascites | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Visceral and Transplantation Surgery, Heidelberg, Germany